CLINICAL TRIAL: NCT06732791
Title: A Comparative Analysis of MGAP and GAP Trauma Scores in Predicting Prognosis for Multiple Trauma Patients: A Prospective Observational Study
Brief Title: Comparative Analysis of MGAP and GAP Trauma Scores in Predicting Outcomes for Multiple Trauma Patients
Acronym: MGAP-GAP
Status: Recruiting | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB20241210B; 010 (Registry Identifier: Nahrain Medical Research Collective (NMRC))
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Trauma
Keywords: MGAP; GAP
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this prospective cohort study is to compare the predictive accuracy of the MGAP and GAP trauma scores in determining the prognosis of multiple trauma patients admitted to the emergency department at Al-Kadhimiya Teaching Hospital, Iraq.

The main questions it aims to answer are:

Does the MGAP score provide a more accurate prediction of outcomes compared to the GAP score? Are there specific subgroups of trauma patients where one score demonstrates superior predictive utility over the other?

Participants will:

Be assessed using both the MGAP and GAP scores upon admission to the emergency department.

Have their clinical outcomes, including mortality, length of stay, and need for surgery, tracked throughout their hospital stay.

DETAILED DESCRIPTION:
Lower-middle income countries (LMICs) pay the price of a growing volume of trauma, as collateral damage for development, rapid urbanization and sociodemographic transition. Trauma includes various types of injuries, which can be either penetrating or non-penetrating, typically categorized as unintentional (like those from road accidents, falls, drownings, and burns) or intentional (including self-inflicted harm and violence). According to the WHO Global Burden of Disease project, around one billion individuals require trauma-related healthcare each year, accounting for 12% of the total global disease burden. Trauma represents a significant global health challenge, causing more fatalities than HIV/AIDS, tuberculosis, malaria, and maternal mortality combined, with over five million deaths annually attributed to traumatic injuries. This makes trauma the fourth leading cause of death worldwide, and the WHO predicts a 40% increase in trauma-related fatalities by 2030, with nearly 90% of these deaths occurring in low and middle-income countries. Most trauma-related deaths happen shortly after the injury occurs, predominantly during the pre-hospital phase, which requires emergency service providers to quickly evaluate the patient's condition and the severity of the trauma to ensure proper referrals.

Research indicates that between 25% and 50% of trauma-related deaths are preventable. The mortality rate serves as the most reliable indicator of trauma prognosis, which can be assessed in two time frames: short-term (within 24 hours) and long-term (over four weeks). An efficient scoring system for trauma patients can assist physicians in rapidly and accurately evaluating injury severity and determining patient management. Timely intervention is crucial in trauma care, as providing swift and suitable treatment has been proven to reduce both mortality and morbidity rates consistently. Such prompt care depends on effective risk stratification in emergency settings. Currently, there are several trauma scoring systems available, each with differing accuracy and reliability for assessing morbidity and mortality risks in patients. Among these are the MGAP and GAP scores, which are simplified, physiologically-based scoring systems not yet widely implemented in low- and middle-income countries. The MGAP acronym stands for "mechanism of injury, GCS, age, and systolic blood pressure," and this score was initially developed in France as a pre-hospital triage tool to predict 30-day mortality. It has also been validated as effective in predicting prolonged ICU stays and major hemorrhages within a European demographic. The MGAP score has been adapted into the GAP score, which omits the injury mechanism for ease of use in clinical environments. GAP stands for "GCS, age, and systolic blood pressure," and it has been validated using data from the Japan Trauma Data Bank. Sartorius et al. determined in their research that the MGAP score can effectively predict the mortality rate of hospitalized trauma patients. Similarly, Yutaka Kondo et al. found that the GAP score can reliably predict the mortality rate of trauma patients in a hospital setting.

Despite advancements in trauma care, predicting outcomes for multiple trauma patients remains a critical challenge in clinical settings, particularly in low-resource environments like Iraq. There is a concerning scarcity of studies within the Iraqi context that evaluate the validity and reliability of scoring systems tailored to the region's unique demographic and healthcare landscape. This underscores the urgent need for comprehensive research to assess the efficacy of the MGAP and GAP Trauma Scores in predicting outcomes for multiple trauma patients in Iraq. Therefore, this study aims to evaluate the effectiveness, reliability, and accuracy of the MGAP and GAP Trauma Scores in assessing the severity of injuries and predicting outcomes for a diverse population of multiple trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 years or older.
* Patients presenting with multiple trauma (Multiple trauma is defined as injuries involving two or more body regions or organ systems that might need coordinated multidisciplinary management).
* Patients presenting to the emergency department within 6 hours of sustaining trauma.
* Patients or their legal representatives must provide informed consent for participation in the study.

Exclusion Criteria:

* Transfers from other facilities with interventions that may affect GAP or MGAP reliability.
* Pregnant women.
* Burn injuries represent the primary mechanism of trauma.
* Incomplete records or failure of follow-up
* Patients who are deceased upon arrival at the emergency department.
* Patient discharge against medical advice.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include patients presenting with multiple trauma to the Trauma and Emergency Department at Al-Kadhimiya Teaching Hospital, Iraq. This population comprises patients who have sustained injuries affecting multiple body regions and require urgent medical evaluation and management
Sampling Method: Non-Probability Sample
Enrollment: 522 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
In hospital mortality | In-Hospital Phase (average of 7-10 days through discharge)
  Mortality (death) during hospitalization.
Accuracy Assessment of the MGAP score | the first 4 hours after ER admission
  (mechanism, Glasgow coma scale, age, and blood pressure), Total scores can range from 3 to 29, with a higher score predicting a better prognosis.
Accuracy Assessment of the GAP score | the first 4 hours after ER admission
  Glasgow coma scale, age, and blood pressure (GAP) score: Total score ranges from 3 to 24. Higher scores suggest a better outcome.

SECONDARY OUTCOMES:
Length of Hospitalization | Up to discharge, an average of 7-10 days
  The total duration of a patient's stay in the hospital, measured from the date of admission to the date of discharge. This includes all days spent in general wards, intensive care units (ICU), and other hospital departments as part of their treatment course.
Need for ICU Admission | Up to discharge, an average of 7-10 days
  The requirement for admission to the intensive care unit (ICU) is determined by the presence of severe clinical deterioration, significant complications, or the need for advanced monitoring and life-support measures.
Need for Surgical Intervention | Up to discharge, an average of 7-10 days
  need for surgical intervention during a trauma patient's hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad A. Hamdawi, Lecturer of general surgery, Study Director — College Of Medicine - Nahrain University
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Result] Kondo Y, Abe T, Kohshi K, Tokuda Y, Cook EF, Kukita I. Revised trauma scoring system to predict in-hospital mortality in the emergency department: Glasgow Coma Scale, Age, and Systolic Blood Pressure score. Crit Care. 2011 Aug 10;15(4):R191. doi: 10.1186/cc10348. PMID 21831280
- [Result] Raux M, Sartorius D, Le Manach Y, David JS, Riou B, Vivien B. What do prehospital trauma scores predict besides mortality? J Trauma. 2011 Sep;71(3):754-9. doi: 10.1097/TA.0b013e3181fd0dae. PMID 21336194
- [Result] Sartorius D, Le Manach Y, David JS, Rancurel E, Smail N, Thicoipe M, Wiel E, Ricard-Hibon A, Berthier F, Gueugniaud PY, Riou B. Mechanism, glasgow coma scale, age, and arterial pressure (MGAP): a new simple prehospital triage score to predict mortality in trauma patients. Crit Care Med. 2010 Mar;38(3):831-7. doi: 10.1097/CCM.0b013e3181cc4a67. PMID 20068467
- [Result] Orhon R, Eren SH, Karadayi S, Korkmaz I, Coskun A, Eren M, Katrancioglu N. Comparison of trauma scores for predicting mortality and morbidity on trauma patients. Ulus Travma Acil Cerrahi Derg. 2014 Jul;20(4):258-64. doi: 10.5505/tjtes.2014.22725. PMID 25135020
- [Result] Nirula R, Maier R, Moore E, Sperry J, Gentilello L. Scoop and run to the trauma center or stay and play at the local hospital: hospital transfer's effect on mortality. J Trauma. 2010 Sep;69(3):595-9; discussion 599-601. doi: 10.1097/TA.0b013e3181ee6e32. PMID 20838131
- [Result] Shoko T, Shiraishi A, Kaji M, Otomo Y. Effect of pre-existing medical conditions on in-hospital mortality: analysis of 20,257 trauma patients in Japan. J Am Coll Surg. 2010 Sep;211(3):338-46. doi: 10.1016/j.jamcollsurg.2010.04.010. Epub 2010 Jul 13. PMID 20800190
- [Result] Rehn M, Perel P, Blackhall K, Lossius HM. Prognostic models for the early care of trauma patients: a systematic review. Scand J Trauma Resusc Emerg Med. 2011 Mar 20;19:17. doi: 10.1186/1757-7241-19-17. PMID 21418599
- [Result] MacKenzie EJ, Rivara FP, Jurkovich GJ, Nathens AB, Frey KP, Egleston BL, Salkever DS, Scharfstein DO. A national evaluation of the effect of trauma-center care on mortality. N Engl J Med. 2006 Jan 26;354(4):366-78. doi: 10.1056/NEJMsa052049. PMID 16436768
- [Result] GBD 2016 Causes of Death Collaborators. Global, regional, and national age-sex specific mortality for 264 causes of death, 1980-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1151-1210. doi: 10.1016/S0140-6736(17)32152-9. PMID 28919116
- [Result] GBD 2013 Mortality and Causes of Death Collaborators. Global, regional, and national age-sex specific all-cause and cause-specific mortality for 240 causes of death, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Jan 10;385(9963):117-71. doi: 10.1016/S0140-6736(14)61682-2. Epub 2014 Dec 18. PMID 25530442
- [Result] Gerdin M, Roy N, Khajanchi M, Kumar V, Fellander-Tsai L, Petzold M, Tomson G, von Schreeb J; Towards Improved Trauma Care Outcomes in India (TITCO). Validation of a novel prediction model for early mortality in adult trauma patients in three public university hospitals in urban India. BMC Emerg Med. 2016 Feb 22;16:15. doi: 10.1186/s12873-016-0079-0. PMID 26905408
- [Result] Haagsma JA, Graetz N, Bolliger I, Naghavi M, Higashi H, Mullany EC, Abera SF, Abraham JP, Adofo K, Alsharif U, Ameh EA, Ammar W, Antonio CA, Barrero LH, Bekele T, Bose D, Brazinova A, Catala-Lopez F, Dandona L, Dandona R, Dargan PI, De Leo D, Degenhardt L, Derrett S, Dharmaratne SD, Driscoll TR, Duan L, Petrovich Ermakov S, Farzadfar F, Feigin VL, Franklin RC, Gabbe B, Gosselin RA, Hafezi-Nejad N, Hamadeh RR, Hijar M, Hu G, Jayaraman SP, Jiang G, Khader YS, Khan EA, Krishnaswami S, Kulkarni C, Lecky FE, Leung R, Lunevicius R, Lyons RA, Majdan M, Mason-Jones AJ, Matzopoulos R, Meaney PA, Mekonnen W, Miller TR, Mock CN, Norman RE, Orozco R, Polinder S, Pourmalek F, Rahimi-Movaghar V, Refaat A, Rojas-Rueda D, Roy N, Schwebel DC, Shaheen A, Shahraz S, Skirbekk V, Soreide K, Soshnikov S, Stein DJ, Sykes BL, Tabb KM, Temesgen AM, Tenkorang EY, Theadom AM, Tran BX, Vasankari TJ, Vavilala MS, Vlassov VV, Woldeyohannes SM, Yip P, Yonemoto N, Younis MZ, Yu C, Murray CJ, Vos T. The global burden of injury: incidence, mortality, disability-adjusted life years and time trends from the Global Burden of Disease study 2013. Inj Prev. 2016 Feb;22(1):3-18. doi: 10.1136/injuryprev-2015-041616. Epub 2015 Dec 3. PMID 26635210
- [Result] Lozano R, Naghavi M, Foreman K, Lim S, Shibuya K, Aboyans V, Abraham J, Adair T, Aggarwal R, Ahn SY, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Barker-Collo S, Bartels DH, Bell ML, Benjamin EJ, Bennett D, Bhalla K, Bikbov B, Bin Abdulhak A, Birbeck G, Blyth F, Bolliger I, Boufous S, Bucello C, Burch M, Burney P, Carapetis J, Chen H, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahodwala N, De Leo D, Degenhardt L, Delossantos A, Denenberg J, Des Jarlais DC, Dharmaratne SD, Dorsey ER, Driscoll T, Duber H, Ebel B, Erwin PJ, Espindola P, Ezzati M, Feigin V, Flaxman AD, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabriel SE, Gakidou E, Gaspari F, Gillum RF, Gonzalez-Medina D, Halasa YA, Haring D, Harrison JE, Havmoeller R, Hay RJ, Hoen B, Hotez PJ, Hoy D, Jacobsen KH, James SL, Jasrasaria R, Jayaraman S, Johns N, Karthikeyan G, Kassebaum N, Keren A, Khoo JP, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lipnick M, Lipshultz SE, Ohno SL, Mabweijano J, MacIntyre MF, Mallinger L, March L, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGrath J, Mensah GA, Merriman TR, Michaud C, Miller M, Miller TR, Mock C, Mocumbi AO, Mokdad AA, Moran A, Mulholland K, Nair MN, Naldi L, Narayan KM, Nasseri K, Norman P, O'Donnell M, Omer SB, Ortblad K, Osborne R, Ozgediz D, Pahari B, Pandian JD, Rivero AP, Padilla RP, Perez-Ruiz F, Perico N, Phillips D, Pierce K, Pope CA 3rd, Porrini E, Pourmalek F, Raju M, Ranganathan D, Rehm JT, Rein DB, Remuzzi G, Rivara FP, Roberts T, De Leon FR, Rosenfeld LC, Rushton L, Sacco RL, Salomon JA, Sampson U, Sanman E, Schwebel DC, Segui-Gomez M, Shepard DS, Singh D, Singleton J, Sliwa K, Smith E, Steer A, Taylor JA, Thomas B, Tleyjeh IM, Towbin JA, Truelsen T, Undurraga EA, Venketasubramanian N, Vijayakumar L, Vos T, Wagner GR, Wang M, Wang W, Watt K, Weinstock MA, Weintraub R, Wilkinson JD, Woolf AD, Wulf S, Yeh PH, Yip P, Zabetian A, Zheng ZJ, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Global and regional mortality from 235 causes of death for 20 age groups in 1990 and 2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2095-128. doi: 10.1016/S0140-6736(12)61728-0. PMID 23245604
- [Result] WHO. World report on Preventing injuries and violence: an overview. Geneva: World Health Organization; 2022.
- [Result] Global Burden of Disease Study 2013 Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 301 acute and chronic diseases and injuries in 188 countries, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Aug 22;386(9995):743-800. doi: 10.1016/S0140-6736(15)60692-4. Epub 2015 Jun 7. PMID 26063472